CLINICAL TRIAL: NCT03052660
Title: Impact of Preoperative Midazolam on Outcome of Elderly Patients: a Multicentre Randomised Controlled Trial
Brief Title: Impact of Preoperative Midazolam on Outcome of Elderly Patients
Acronym: I-PROMOTE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-115
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Preanesthetic Medication
Keywords: Midazolam; Anxiety; Clinical trial; Patient Satisfaction
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam (Experimental): Midazolam, 3.75 mg , oral, once, 30-45 minutes before surgery
  Interventions: Drug: Midazolam
- Placebo (Placebo Comparator): Placebo, oral, once, 30-45 minutes before surgery
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Midazolam — Oral administration preoperatively
  Other Names: Dormicum
  Arms: Midazolam
Drug: Placebo oral capsule — Oral administration preoperatively
  Arms: Placebo

SUMMARY:
We aim to assess, if placebo compared to preoperative administration of midazolam in elderly patients is equal in regard to the global postoperative patient satisfaction

DETAILED DESCRIPTION:
Generalised premedication with benzodiazepines in all surgical patients has become questionable, regarding the risk-benefit assessment and the lack of evidence for this practice. Particularly, in elderly patients (≥65 years), a higher risk for adverse events is described.

Patients will be randomly assigned to one of the following two study groups. Preoperatively, group 1 will receive midazolam and group 2 will receive placebo.

Anaesthesia will be performed according to the clinical routine.

All possible side effects are described in the SmPC for midazolam. For the placebo-group, we do not expect any harm, as in the case of strong preoperative anxiety or agitation, additional midazolam application may occur on behalf of the attending anaesthesist at any time.

The sample size was calculated based on detecting a minimum of 5 unit difference in the primary outcome variable overall patient satisfaction measured with the EVAN-G. Setting a type 1 error of 0.05, a power of 0.8 and assuming the standard deviation of EVAN-G to be 14 units, 248 patients per group are needed to detect a 5 unit difference.

Considering a drop-out of 10% and a screening failure of 10%, we decided to include 614 patients in total.

The hypothesis of the study is that global patient satisfaction after surgery in elderly patients is similar after preoperative placebo application compared to midazolam application.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Only legally competent patients
2. Written informed consent prior to study participation
3. 65-80 years
4. Elective surgery
5. Expected surgery duration ≥ 30 minutes
6. Planned general or combined regional and general anaesthesia
7. Planned extubation at the end of surgery

Exclusion Criteria:

1. Age > 80 years
2. Age < 65 years
3. Non-fluency in German language
4. Alcohol and/ or drugs abuse
5. Chronic benzodiazepine treatment
6. Intracranial surgery
7. Local and stand by anaesthesia or solely regional anaesthesia
8. Monitored anaesthesia care
9. Cardiac surgery
10. Ambulatory surgery
11. Repeated surgery
12. Contraindications for benzodiazepine application (e.g. sleep apnoea syndrome, severe chronic obstructive pulmonary disease, allergy)
13. Allergy against any component of the Placebo (lactose monohydrate, cellulose powder, magnesium stearate, microcrystalline cellulose) or investigational drug (midazolam, lactose) or the capsules (gelatine, E171 titanium dioxide, E132 indigotine).
14. Expected benzodiazepine requirement after surgery
15. Expected continuous mandatory ventilation after surgery
16. Patients who explicitly request anxiolytic premedication
17. Patients with severe neurological or psychiatric disorders
18. Refusal of study participation by the patient
19. Parallel participation in interventional clinical studies within the last 30 days

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 782 (Actual)
Dates: Start 2017-10-12 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Global patient satisfaction on the first postoperative day | on the first postoperative day (1 day)
  measured with the EVAN-G questionnaire on the first postoperative day

SECONDARY OUTCOMES:
Cognitive testing | preoperative, day 1 and day 30 after surgery (31 days)
  Measured by the short blessed test
Delirium testing | preoperative, day 1 after surgery (2 days)
  Measured by Confusion Assessment Method (CAM)
Preoperative anxiety | preoperatively (1 day)
  Measured by Amsterdam Preoperative Anxiety and Information Scale (APAIS)
Change of health-related quality of life | preoperative and day 30 after surgery (31 days)
  Measured by the individual health-related quality of life assessment EQ-5D-5L
Activities of daily living | preoperative and day 30 after surgery (31 days)
  Measured by Instrumental Activities of Daily Living scale (IADL)
Perception of pain, well-being, and sleeping | preoperative until first postoperative day (3 days)
  Self-reported by visual analogue scale (VAS)
Number of participants with adverse events and serious adverse events | surgery and first postoperative day (2 days)
  Review of medical charts and patient interview
Patient cooperation | surgery day (1 day)
  Self-reported by visual analogue scale (VAS) by the attending anesthetist
Anaesthesia related data | surgery day (1 day)
  Anesthesia drugs, type of anesthesia, duration, extubation-time
Surgery related data | surgery day (1 day)
  Duration and kind of surgery
Rescue benzodiazepine application | surgery day (1 day)
  assessment of additional requirement of midazolam in the operating area
Patients vital data | surgery day (1 day)
  Measurement of SpO2, RRsys, HR on arrival in the operating room and at the end of surgery
Mortality | 30 days
  Patient chart review and telephone interview after discharge
Major adverse events | 30 days
  Assessment of postoperative major adverse cardiovascular and cerebral events by patient chart review and telephone interview after discharge
Hospital length of stay | on postoperative day 30 (1 day)
  Patient chart review
Intensive care unit length of stay | on postoperative day 30 (1 day)
  Patient chart review

CONTACTS AND LOCATIONS:
Overall Officials: Mark Coburn, Professor, Study Chair — Department of Anesthesiology, University Hospital Aachen, Germany
Locations (9):
- Germany (9):
  - Department of Anesthesiology, University Hospital Aachen, Aachen, North Rhine-Westphalia
  - Klinik für Anästhesiologie und Operative Intensivmedizin, Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Klinik für Anästhesiologie, Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Marien-Hospital Herne, Herne
  - Universitätsklinikum Magdeburg A.ö.R., Magdeburg
  - Department of Anaesthesiology, University Hospital Klinikum rechts der Isar Munich, Munich
  - LMU München, München
  - Kreiskliniken Reutlingen, Klinikum am steinenberg, Reutlingen
  - Klinik für Anästhesiologie und Intensivmedizin, Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Auquier P, Pernoud N, Bruder N, Simeoni MC, Auffray JP, Colavolpe C, Francois G, Gouin F, Manelli JC, Martin C, Sapin C, Blache JL. Development and validation of a perioperative satisfaction questionnaire. Anesthesiology. 2005 Jun;102(6):1116-23. doi: 10.1097/00000542-200506000-00010. PMID 15915023
- [Result] American Geriatrics Society Expert Panel on Postoperative Delirium in Older Adults. American Geriatrics Society abstracted clinical practice guideline for postoperative delirium in older adults. J Am Geriatr Soc. 2015 Jan;63(1):142-50. doi: 10.1111/jgs.13281. Epub 2014 Dec 12. PMID 25495432
- [Result] Maurice-Szamburski A, Auquier P, Viarre-Oreal V, Cuvillon P, Carles M, Ripart J, Honore S, Triglia T, Loundou A, Leone M, Bruder N; PremedX Study Investigators. Effect of sedative premedication on patient experience after general anesthesia: a randomized clinical trial. JAMA. 2015 Mar 3;313(9):916-25. doi: 10.1001/jama.2015.1108. PMID 25734733
- [Derived] Kowark A, Keszei AP, Schneider G, Pilge S, Schneider F, Obert DP, Georgii MT, Heim M, Rossaint R, Ziemann S, van Waesberghe J, Czaplik M, Puhringer FK, Minarski C, May V, Malisi T, Drexler B, Ring CM, Engler P, Tilly R, Bischoff P, Frey U, Wittmann M, Soehle M, Saller T, Kienbaum P, Kretzschmar M, Coburn M; I-PROMOTE Study Group. Preoperative Midazolam and Patient-Centered Outcomes of Older Patients: The I-PROMOTE Randomized Clinical Trial. JAMA Surg. 2024 Feb 1;159(2):129-138. doi: 10.1001/jamasurg.2023.6479. PMID 38117527
- [Derived] Wang ML, Min J, Sands LP, Leung JM; the Perioperative Medicine Research Group. Midazolam Premedication Immediately Before Surgery Is Not Associated With Early Postoperative Delirium. Anesth Analg. 2021 Sep 1;133(3):765-771. doi: 10.1213/ANE.0000000000005482. PMID 33721875
- [Derived] Kowark A, Rossaint R, Keszei AP, Bischoff P, Czaplik M, Drexler B, Kienbaum P, Kretzschmar M, Rex C, Saller T, Schneider G, Soehle M, Coburn M; I-PROMOTE study group. Impact of PReOperative Midazolam on OuTcome of Elderly patients (I-PROMOTE): study protocol for a multicentre randomised controlled trial. Trials. 2019 Jul 15;20(1):430. doi: 10.1186/s13063-019-3512-3. PMID 31307505